CLINICAL TRIAL: NCT06867692
Title: Effects of Aerobic Exercises on Dual-task Performance and Motor Skills in Children With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/G-III/RCR&AHS/B42-176
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment
Keywords: Mild Cognitive Impairment; Dual-task performance; Aerobic exercises
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light Physical Activity Plan (Experimental)
  Interventions: Other: Light Physical Activity Plan
- Aerobic Exercise (Active Comparator)
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Warm-Up (5 minutes): Marching in Place: 2 minutes of marching to elevate heart rate. Arm Circles: 1 minute of small and large arm circles. Side Steps with Arm Swings: 2 minutes of stepping side to side with gentle arm swings. Main Exercise Routine (35 minutes): Walking/Jogging Intervals: 10 minutes alternating between 1 minute of walking and 1 minute of jogging. Jumping rope: 10 minutes of rope jumping. As a pre-determined routine to maintain consistency. Aerobic Games: 10 minutes of structured games like:
  1. Simon Says: Incorporating aerobic movements like jumping jacks, running in place, etc.
  2. Obstacle Course: Pre-planned course involving stepping over objects, crawling, and balancing. Ball Activities: 5 minutes of activities such as throwing and catching, or dribbling a ball around cones.
  3. Cool Down (5 minutes) Stretching: Gentle stretching of major muscle groups, holding each stretch for 20-30 seconds.
  Arms: Aerobic Exercise
Other: Light Physical Activity Plan — Warm-Up (5 minutes): Gentle Walking: 2 minutes at a slow pace. Light Arm Movements: 1 minute of gently moving arms up and down. Side Steps: 2 minutes of gentle side stepping.
  2. Main Activity Routine (35 minutes): Stretching Exercises: 10 minutes of gentle stretching, focusing on flexibility. Balance Activities: 10 minutes of activities such as: Standing on One Leg: Holding balance for 10-15 seconds on each leg. Heel-to-Toe Walking: Walking in a straight line, placing the heel of one foot directly in front of the toes of the other foot. 3. Light Coordination Games: 10 minutes of low-intensity activities like: Passing a Ball: Gently passing a ball back and forth with a partner. Basic Catch and Throw: Simple throw and catch exercises with a soft ball. Guided Relaxation: 5 minutes of guided relaxation techniques, including deep breathing and visualization. 4. Cool Down (5 minutes) Gentle Stretching: Stretching major muscle groups, holding each stretch for 20-30 second
  Arms: Light Physical Activity Plan

SUMMARY:
Cognition refers to the mental processes involved in gaining knowledge and understanding, encompassing aspects such as thinking, knowing, remembering, judging, and problem-solving. These processes include attention, memory, executive functions, perception, language, and visuospatial skills. In children, cognitive development is critical for academic success, social interactions, and daily living activities. In the context of mild cognitive impairment (MCI) in children, cognitive processes may be less efficient or slower than in typically developing peers.This can affect their ability to perform tasks that require simultaneous cognitive and motor functions, known as dual tasks. Aerobic exercises are known to provide numerous cognitive and physical benefits, but their specific impact on children with MCI has not been thoroughly investigated. The aim of study is to analyze the effects of aerobic exercises on dual-task performance and motor skills in children with mild cognitive impairment.The current study will be randomized control trial; data will be collected from Government special education center Johar Town. The study will include patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will be both genders, having age between7 to 12, children with IQ ranging from 50-70, who are cooperative. Children with Hearing or vision impairment, any neurological/musculoskeletal disorder or already involved in an intervention program will also be excluded from the study. Experimental group will perform a structured aerobic exercise program and control group will do its daily routine activities. The intervention group will receive 3 sessions per week for 12weeks. Each session lasted 45 min on average. Outcomes to be analyzed will be dual-task performance and motor skills. Tools used for data collection will be Timed Up and Go, Single Leg Stance, Tandem Stance, and 30-second Sit-to-Stand tests and TGMD-2. Data will be analyzed through SPSS version 26.00.

ELIGIBILITY:
Inclusion Criteria:

* IQ from 50 to 70
* Who can easily understand instructions
* Both genders are included

Exclusion Criteria:

* Hearing or vision impairment
* Any neurological/musculoskeletal disorder
* Already involved in an intervention program

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go | Baseline and 12th week
  In this test, the child wears their usual footwear and is instructed to stand up from a chair, walk a designated distance of 3 meters at a comfortable and safe pace, turn around, walk back to the chair, and sit down. The time taken to complete the task 10 is recorded in seconds using a stopwatch.
Single Leg Stance | Baseline and 12th week
  During the test, the child is instructed to lift one leg and stand unassisted, maintaining this position for as long as possible. The duration until the foot touches the ground is timed in seconds using a stopwatch.
Tandem Stance | Baseline and 12th week
  In the Tandem Stance test, the child is asked to stand with one foot directly in front of the other in a heel-to-toe position, thereby narrowing the base of support to assess static balance. The test ends when the child can no longer maintain this position, and the duration is timed in seconds using a stopwatch. If the child can hold the tandem stance for 30 seconds, the test is not repeated.
30-second Sit-to-Stand tests | Baseline and 12th week
  In this test, the child is instructed to stand up from a chair (seat height 43 cm) with a straight back and no armrests, keeping their arms crossed over their chest, then sit back down and repeat this for 30 seconds. The number of times the child stands up in 30 seconds is recorded.
TGMD-2 | Baseline and 12th week
  The TGMD-2 (Test of Gross Motor Development, Second Edition) is a widely used assessment tool designed to evaluate the gross motor skills of children. It assesses both locomotor (movement from one place to another) and object control (handling and manipulation of objects) skills.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Hands on Care, Wapda Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen CY, Lawlor JP, Duggan AK, Hardy JB, Eaton WW. Mild cognitive impairment in early life and mental health problems in adulthood. Am J Public Health. 2006 Oct;96(10):1772-8. doi: 10.2105/AJPH.2004.057075. PMID 17008572
- [Background] Vuijk PJ, Hartman E, Scherder E, Visscher C. Motor performance of children with mild intellectual disability and borderline intellectual functioning. J Intellect Disabil Res. 2010 Nov;54(11):955-65. doi: 10.1111/j.1365-2788.2010.01318.x. Epub 2010 Sep 20. PMID 20854287
- [Background] Buyukcelik NM, Yigit S, Turhan B. An investigation of the effects of dual-task balance exercises on balance, functional status and dual-task performance in children with Down syndrome. Dev Neurorehabil. 2023 Jul;26(5):320-327. doi: 10.1080/17518423.2023.2233031. Epub 2023 Jul 4. PMID 37403442